CLINICAL TRIAL: NCT04371146
Title: The Role of Dopaminergic and Noradrenergic Neurotransmission in Value- and Salience-based Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Value-Salience-2017-0444
Record Dates: First submitted 2020-04-26; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Methylphenidate; Reboxetine

STUDY DESIGN:
Intervention Model Description: The investigators implement a randomized, double-blind, placebo-controlled between-subjects design, using one factor (pharmacological intervention) with three levels (reboxetine, methylphenidate and placebo).
Who Masked: Participant, Investigator
Masking Description: All participants will receive the same instructions, and neither the participants nor the experimenters are informed which drug is used. Participants must take the drug in front of the investigator, to ensure correct intake and compliance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dopamine reuptake inhibitor (Experimental): Participants in the dopamine reuptake inhibitor group will be asked to take one pill containing 35 mg methylphenidate 1.5 hours before performing the tasks.
  Interventions: Drug: Methylphenidate
- Noradrenaline reuptake inhibitor (Experimental): Participants in the noradrenaline reuptake inhibitor group will be asked to take one pill containing 8 mg reboxetine 1.5 hours before performing the tasks.
  Interventions: Drug: Reboxetine
- Placebo (Placebo Comparator): Participants in the placebo group will be asked to take a placebo pill 1.5 hours before performing the tasks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Methylphenidate — 35 mg methylphenidate (Ritalin®) is administered once using a randomized placebo-controlled between subject's design
  Other Names: Ritalin®
  Arms: Dopamine reuptake inhibitor
Drug: Reboxetine — 8 mg Reboxetine (Edronax®) is administered once using a randomized placebo-controlled between subject's design
  Other Names: Edronax®
  Arms: Noradrenaline reuptake inhibitor
Drug: Placebos — A placebo pill is administered once using a randomized placebo-controlled between subject's design
  Other Names: Placebo Pill
  Arms: Placebo

SUMMARY:
Approach versus avoidance decisions are at the centre of adaptive behaviour and survival. These decisions are thought to be guided by the value of the choice options, which are a function of the magnitude of predicted rewards and punishments. Moreover, the allocation of attention to choice options is thought to be driven by salience, i.e. the overall importance of the predicted outcomes. While salience increases with the magnitude of both predicted rewards and predicted punishments, value increases with reward but decreases with punishment. In previous research, value and salience have often remained confounded during value-based decision making. Rodent research suggests that value is associated with dopamine and salience with norepinephrine. The present study aims at disentangling value from salience processing during decision-making tasks in healthy subjects by administering dopamine or noradrenaline reuptake inhibitors. This is done by using a single dose challenge in a randomized placebo-controlled between subject's design, administering either methylphenidate (35 mg), reboxetine (8 mg), or placebo to healthy young participants before they perform tasks tapping into various aspects of value and salience.

ELIGIBILITY:
Inclusion Criteria:

* Physically and psychiatrically healthy men and women aged ≥ 18- ≤ 35 years
* Ability and willingness to participate in the study
* Signed informed consent

Exclusion Criteria:

* Serious past brain disease or injury (data quality)
* Frequent headaches (of any sort, > 1/week) or migraine (irrespective of frequency)
* History of epileptic seizures
* Any neurological disorder
* Surgery to head or heart (safety, potential metal pieces)
* Pacemaker, hearing aid or neurostimulator (safety, metal pieces)
* Known cardiac or cardiovascular disease or anomaly
* Family history of sudden death due to cardiac arrhythmia
* High or low blood pressure, history of heart attack, infrequent heartbeat
* Respiratory problems (including difficulty with breathing through the nose)
* Glaucoma (present or in history)
* Insufficiency of kidney or liver, acute liver disease
* Any psychiatric disorder (especially depression, mania, schizophrenia, addiction and suicidality)
* Severe vocal or motor tics (methylphenidate, data quality)
* Severe psychosomatic disorder (somatic complaints without clear medical cause, has a mental component)
* Pregnancy, nursing, or currently planned pregnancy
* Current allergy in general or allergy to methylphenidate or reboxetine
* Severe intolerance to lactose including strong diarrhea after only a few mg (weak lactose intolerance is no exclusion criterion as medication only contains slightest dosage (around 4mg) of lactose)
* Currently taking any medication that might interfere with Methylphenidate and Reboxetine, especially MAO-Inhibitors (e.g. Aurorix (Moclobemid) und Azilect (Rasagilin), antipsychotics, antibiotics, and medication for heart diseases
* Currently taking any further medication (besides birth control) or natural products (infrequent intake of natural products and/or food supplements need to be mentioned to the examiner)
* Drug abuse (current or past abuse; in case of single use please inform the examiner)
* Serious acute or chronic disease that could interfere with participation in the experiments
* Inability to understand the instructions or insufficient comprehension of German language
* Participants having their weight outside of the range of ≥ 60 kg - ≤ 80 kg
* Clinically relevant score in STAI T (anxiety), measured during prescreening on a separate day
* Long QT syndrome or other arrhythmias, measured during prescreening on a separate day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Response time data | These tasks take place 1,5 hours after the drug was administered
  The investigators record responses and specifically reaction times during 5 different decision-making tasks.
  In a value vs salience task, value and salience processing is disentangled during value-based decision-making. Participants either accept or reject compound stimuli that were before associated with monetary outcomes.
  In a face in the crowd task, participants detect a target face (angry vs happy) in a crowd of opposite face type.
  During a task on risk and ambiguity decision-making, participants have to decide between safe and lottery options associated with either monetary risk or ambiguity.
  In an adaptive risk-taking task, participants have to choose between two risky monetary options.
  In an effort task, participants decide whether they are willing to exert physical effort for monetary reward.
  Response times are measured in milliseconds from the tasks. The investigators calculate how long participants take to make decisions in each trial.
Choice data | These tasks take place 1,5 hours after the drug was administered
  As a dependent variable the investigators record responses and specifically choices made during the above-mentioned different decision-making tasks. The investigators evaluate what kind of answers were made during each trial of the decision-making tasks, in respect to correctness or preference (percentage).

SECONDARY OUTCOMES:
Computational modelling applied to choice data | These tasks take place 1,5 hours after the drug was administered
  Computational parameters are mathematically estimated from the data of participants during the above-mentioned decision-making tasks. Specifically, mathematical models will be applied to choice data (percentage).
Computational modelling applied to response time data | These tasks take place 1,5 hours after the drug was administered
  Computational parameters are mathematically estimated from the data of participants during the above-mentioned decision-making tasks. Specifically, mathematical models will be applied to response time data (milliseconds).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Tobler, PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland